CLINICAL TRIAL: NCT01652989
Title: 5-Year Controlled Intervention Trial: Testing DVD Versus Group Delivery of a Weight-Loss Maintenance Intervention in Native Hawaiian- Serving Worksites
Brief Title: PILI at Work a 5-Year Controlled Intervention Trial: Testing DVD Versus Group Delivery of a Weight-Loss Maintenance Intervention in Native Hawaiian- Serving Worksites
Acronym: P@W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Queen's Medical Center (Other); I Ola Lahui, Inc. (Other); Queen Lili'uokalani Children's Center (Unknown); Ke Ola Mamo (Other); Molokai Community Health Center (Unknown); Keiki o ka Aina (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U54CA153459 (NIH)
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Overweight; Weight Loss; Weight Loss Maintenance
Keywords: weight loss; weight loss maintenance; community based participatory research; overweight
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight loss maintenance intervention delivered via DVD (Experimental): Weight loss maintenance intervention delivered via DVD (without a peer facilitator) to employee participants within the respective worksites randomized to this arm. Using DVD technology, a total of 11 additional sessions (designed for weight loss maintenance) over a 9-month period will be delivered to the participants of this arm using DVD-produced lessons of PILI Maintenance
  Interventions: Behavioral: Weight loss maintenance intervention delivered via DVD
- Weight loss maintenance intervention Face-to-Face (Experimental): The PILI Maintenance delivered face-to-face in a group setting by trained peer facilitators to employee participants within the respective worksites randomized to this arm. The trained peer facilitator will deliver a total of 11 additional sessions (designed for weight loss maintenance) over a 9-month period, meeting bi-weekly for the first 2 months and then monthly for the remaining 7 months with a group of 8 to 15 participants.
  Interventions: Behavioral: Weight loss maintenance intervention face-to-face

INTERVENTIONS:
Behavioral: Weight loss maintenance intervention face-to-face
  Arms: Weight loss maintenance intervention Face-to-Face
Behavioral: Weight loss maintenance intervention delivered via DVD
  Arms: Weight loss maintenance intervention delivered via DVD

SUMMARY:
The PILI @ Work project is a 5 year randomized control trial to adapt a weight loss program for the employees of Native Hawaiian-serving organizations in Hawai'i. The study has two specific aims:

Specific Aim 1: To adapt and implement a weight loss and weight loss maintenance program in Native Hawaiian-serving organizations, working with employee representatives to determine how the intervention can be best implemented with employees at the worksites. Specific Aim 2: Among employees participating in the program, to test whether weight loss maintenance program in DVD format is as effective as the weight loss maintenance program in a group face to face format in maintaining weight loss for employees who complete weight loss program.

The investigators hypothesize that the PILI @ Work interventions can be effectively adapted and implemented in a worksite settings with active participation by employees and employers. The investigators also hypothesize that overweight (BMI ≥ 25) and obese (BMI ≥ 30) employees who complete weight loss portion of the intervention, and are randomized to received the weight loss maintenance intervention via DVD will have similar success at maintaining weight loss compared to those randomized to PILI Maintenance in group meetings or settings. The investigators hypothesize that will will also be true for physical functioning,blood pressure, daily self-weighing, low to moderate fat and low calorie diets, and daily physical activity.

DETAILED DESCRIPTION:
Effective and culturally relevant interventions are needed to curb the rising tide of overweight and obesity. This study adapts an evidence-based weight loss intervention for use in Native Hawaiian-serving organizations in Hawai'i, using a community-based participatory research (CBPR) approach. Findings from our two previous NIH-funded projects help to inform this proposed research: 1) The Designing Healthy Worksites (DHW) Project and 2) the PILI Lifestyle Intervention (PILI), developed by the PILI 'Ohana (family) Project: Partnerships to Overcome Obesity Disparities in Hawai'i.

The DHW Project engaged with eight Native Hawaiian-serving organizations to obtain data on 1) existing worksite policies that support and/or promote health and well-being of employees and 2) the perspectives and ideas of employees and employers around creating a healthy workplace. DHW participants expressed enthusiasm for health promotion programs at the worksite, especially weight-loss programs.

The PILI 'Ohana Project adapted an evidence-based lifestyle intervention for use with Native Hawaiians and Pacific Islanders who sought care at community health clinics and/or were members of civic groups. The PILI Lifestyle Intervention (PILI) has two phases-PILI Weight Loss and PILI Maintenance. Both PILI Wt Loss and PILI Maintenance were designed for deliver to community-based groups. In pilot testing, all participants participating in PILI Wt Loss and realized significant weight loss after 3 months. Participants then were randomized into PILI Maintenance or standard behavioral treatment (SBT); those in PILI Maintenance performed better than those in SBT. PILI Wt Loss and PILI Maintenance were improved based on feedback from the pilot. Because of reported time constraints by pilot participants, a DVD version of PILI Maintenance was developed that people could use instead of attending group sessions. In a subsequent community-based study of PILI (funded by NIH-NCMHD and now underway), non-worksite participants are being randomized into a face-to-face or DVD delivery of PILI Maintenance after completion of PILI Wt Loss.

Our specific aims and hypotheses for its application in worksites are as follows:

Specific Aim 1: To adapt and implement PILI Wt Loss and PILI Maintenance in Native Hawaiian-serving organizations, working with employee representatives to determine how the intervention can be best implemented with employees in worksites (PILI Wt Loss and PILI Maintenance together will be called PILI@Work).

Primary hypothesis: A community-tested, evidence-based intervention for obesity reduction and weight-loss maintenance can be effectively adapted and implemented in worksite settings with active participation by employees and employers.

Specific Aim 2: Among employees participating in PILI@Work, to test whether PILI Maintenance in DVD format is as effective as PILI Maintenance in Group in maintaining weight loss for employees who complete PILI Wt Loss.

Primary hypothesis: Overweight (BMI ≥ 25) and obese (BMI ≥ 30) employees who complete PILI Wt Loss will have successful weight loss outcomes, and those randomized to PILI Maintenance in DVD will have similar success at maintaining weight loss compared to those randomized to PILI Maintenance in group meetings or settings. Successful weight loss maintenance will be measured as a ≥ 3% mean weight change.

Secondary hypothesis: Employees participating in PILI Maintenance in DVD and those in PILI Maintenance in Group will show similar maintenance of, or improvements in, physical functioning, blood pressure, daily self-weighing, low to moderate fat and low calorie diets, and daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

* persons of any self-reported ethnicity
* age 18 years or older
* overweight or obese as defined as (BMI) ≥ 25 for Caucasians, NHs, or PIs and > 23 for those with Asian ancestry
* willing and able to follow a healthy eating and physical activity regimen that could include 150 minutes of brisk walking per week (or equivalent) and caloric intake control

Exclusion Criteria:

* prognosed survival < 6 months
* planning to terminate employment during the intervention study period (12 months)
* pregnancy
* any dietary or exercise restrictions that would prevent an individual from fully participating in the intervention protocol (e.g., end-stage renal disease on a renal diet)
* any co-morbid condition (physical and mental disabilities) that would prevent the individual from participating in the intervention protocol (e.g., severe arthritis, hemi-paresis, major psychiatric illness, eating disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline to 3-month and 12-month follow up | baseline, 3-months, 12-months
  Change in weight from baseline to 3-month and 12-month follow up.
Change in physical functioning from baseline to 3-month and 12-month follow up | baseline, 3-months, 12-months
  Change in number of feet walked in 6 minutes from baseline to 3-month and 12-month follow up.

SECONDARY OUTCOMES:
Blood pressure | baseline, 3-months, 12-months
  Change in blood pressure from baseline to 3-month and 12-month follow up.
Physical Activity Frequency | baseline, 3-months, 12-month
  Change in physical activity frequency from baseline to 3-month and 12-month follow up as measured by a brief 3-item questionnaire assessing frequency of moderate and vigorous physical activity over the last month.
Fat in Diet | baseline, 3-months, 12-months
  Change in fat in diet from baseline to 3-month and 12-month follow up as measured by a 36-item questionnaire designed to measure the amount of fat in a participant's diet.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Principal Investigator — University of Hawaii at Manoa
Locations (8):
- United States (8):
  - I Ola Lahui, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, John A Burns School of Medicine, Honolulu, Hawaii
  - Ke Ola Mamo, Native Hawaiian Health Care System, Honolulu, Hawaii
  - Queen Liliuokalani Children's Center, Honolulu, Hawaii
  - Keiki o ka Aina, Honolulu, Hawaii
  - Queen Liliuokalani Children's Center, Kailua-Kona, Hawaii
  - Molokai Community Health Center, Kaunakakai, Hawaii